CLINICAL TRIAL: NCT00150423
Title: An Open-Label, Extension Safety and Efficacy Study of Pregabalin in Patients With Painful Diabetic Peripheral Neuropathy.
Brief Title: To Evaluate the Safety and Efficacy of Pregabalin in Patients With Painful Diabetic Peripheral Neuropathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-165
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-01-01 (Estimated); Status verified 2006-12

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate the safety and efficacy of pregabalin in patients with painful diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for the preceding double-blind BID study in painful diabetic peripheral neuropathy
* Must have received pregabalin/placebo under double-blind conditions for a minimum of 3 weeks.

Exclusion Criteria:

* Patients may not participate if they experienced a serious adverse event during the preceding double-blind BID study which was determined to be related to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384
Dates: Start 2001-01; Study Completion 2005-07

PRIMARY OUTCOMES:
Safety Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer